CLINICAL TRIAL: NCT01087138
Title: Effect of Exercise and Calcium Foods on Pubertal Bone Gain
Brief Title: Study to Determine How Exercise and Calcium Affect Pubertal Bone
Acronym: Exkids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Joan M. Lappe, Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 97-11384
Record Dates: First submitted 2010-03-12; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Bone Health
Keywords: bone health; bone density; bone mass
MeSH Terms: interventions — Exercise; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise (Experimental): exercise class 3x's/week
  Interventions: Behavioral: exercise
- exercise and calcium intake (Experimental): exercise class 3x's/week and 1500mg calcium/day
  Interventions: Behavioral: exercise and calcium
- usual exercise and calcium (No Intervention): usual exercise and calcium intake

INTERVENTIONS:
Behavioral: exercise — exercise class 3x's/week
  Arms: Exercise
Behavioral: exercise and calcium — exercise class 3x's/week and 1500mg calcium intake
  Arms: exercise and calcium intake

SUMMARY:
To determine if increasing the amount of calcium that girls eat or the degree of exercise in which they participate will increase their bone strength.

ELIGIBILITY:
Inclusion Criteria:

* 9-10 years of age
* Premenarcheal
* Female

Exclusion Criteria:

* corticosteroid or anticonvulsant therapy
* lactose intolerance or milk allergy
* family history of hypercholesterolemia
* mental or physical handicaps
* chronic disease
* body mass index ³ 85th percentile for age and gender
* baseline calcium intake of > 1100 mg/day
* participation in team sports > 3 times per week

Ages: 9 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Creighton University, Omaha, Nebraska, United States